CLINICAL TRIAL: NCT04987489
Title: A Phase 2 Open-Label Study to Evaluate Safety and Clinical Activity of Etavopivat in Patients With Thalassemia or Sickle Cell Disease
Brief Title: A Study of Etavopivat in Patients With Thalassemia or Sickle Cell Disease
Acronym: GLADIOLUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4202-HEM-201
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease; Thalassemia
Keywords: SCD; sickle cell disease; sickle cell; anemia; sickle cell anemia; hemolytic; hemoglobin; vaso-occlusive crisis; VOC; vaso-occlusive events; sickle cell crisis; pain crisis; pain episode; congenital anemia; hemolytic anemia; hematologic disease; hemoglobinopathy; hemoglobinopathies; genetic disease; inborn disease; sickle cell trait; pyruvate kinase; PKR; thalassemia; beta-thalassemia; alpha-thalassemia; transfusions; hemoglobin H; transfusion; transfusion-dependent; non-transfusion dependent; hemoglobin E
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia; Hemolysis; Vaso-Occlusive Crises; Anemia, Hemolytic; Hematologic Diseases; Hemoglobinopathies; Genetic Diseases, Inborn; Sickle Cell Trait; beta-Thalassemia; alpha-Thalassemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Etavopivat 400 mg daily - SCD with transfusions (Experimental): Patients with sickle cell disease on chronic red blood cell transfusions
  Interventions: Drug: Etavopivat tablets
- Etavopivat 400 mg daily - Thalassemia with transfusions (Experimental): Patients with thalassemia on chronic red blood cell transfusions
  Interventions: Drug: Etavopivat tablets
- Etavopivat 400 mg daily - Thalassemia (Experimental): Patients with thalassemia not on chronic red blood cell transfusions
  Interventions: Drug: Etavopivat tablets

INTERVENTIONS:
Drug: Etavopivat tablets — Etavopivat 400 mg once daily
  Other Names: FT-4202

SUMMARY:
This clinical trial is a Phase 2 study that will evaluate the safety and clinical activity of etavopivat in patients with thalassemia or sickle cell disease and test how well etavopivat works to lower the number of red blood cell transfusions required and increase hemoglobin.

DETAILED DESCRIPTION:
Etavopivat is a potent, selective, orally bioavailable, small-molecule activator of pyruvate kinase red blood cell (PKR) being developed by Forma Therapeutics, Inc and is intended for use as a treatment for patients with sickle cell disease (SCD) or other inherited hemoglobinopathies or refractory anemias. This study is a multicenter, Phase 2, open-label, multiple-cohort study examining the safety and efficacy of etavopivat for the treatment of patients, age 12 to 65 years, with SCD or thalassemia. Three treatment cohorts based on the patients hemoglobinopathy (SCD or thalassemia) and transfusion requirements will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provision of consent
* Female patients of childbearing potential must use acceptable methods of contraception, male patients are willing to use barrier methods of contraception

Cohort A (Sickle Cell Disease Transfusion Cohort)

* Confirmed diagnosis of sickle cell disease
* Chronically red blood cell transfused (sample or exchange [manual or via electrophoresis]) for primary stroke prevention or due to previous stroke. Chronic red blood cell transfusion is defined as: ≥ 6 red blood cell units in the previous 24 weeks before the first dose of study treatment and no transfusion-free period for > 35 days during that period
* At least 24 months of chronic monthly red blood cell transfusions for secondary stroke prevention/treatment of primary stroke (initial completed overt clinical stroke with documented infarction on brain computed tomography [CT] or magnetic resonance imaging [MRI])
* Prior to screening OR at least 12 months of chronic RBC transfusions for primary stroke prevention (abnormal TCD) prior to screening
* Documented adequate monthly transfusions with average HbS ≤ 45% (the upper limit of the established academic community standard) for the previous 12 weeks of red blood cell transfusions before the first dose of study treatment

Cohort B (Thalassemia Transfusion Cohort)

* Documented diagnosis of β-thalassemia, Hemoglobin E/ β-thalassemia or Hemoglobin H (α-thalassemia), or other thalassemia variant
* Chronically transfused, defined as: ≥ 6 red blood cell units in the previous 24 weeks before the first dose of study treatment and no transfusion-free period for > 35 days during that period

Cohort C (Thalassemia Non-transfused Cohort)

* Documented diagnosis of β-thalassemia, Hemoglobin E/ β-thalassemia or Hemoglobin H (α-thalassemia), or other thalassemia variant
* Hemoglobin ≤ 10 g/dL

Exclusion Criteria:

* Female who is breast feeding or pregnant
* Hepatic dysfunction characterized by:

  * Alanine aminotransferase (ALT) > 4.0 × upper limit of normal (ULN)
  * Direct bilirubin > 3.0 × ULN
  * History of cirrhosis
* Known human immunodeficiency virus (HIV) positivity
* Active hepatitis B or hepatitis C infection
* Severe renal dysfunction or on chronic dialysis
* History of malignancy within the past 2 years prior to treatment Day 1 requiring systemic chemotherapy and/or radiation.

  * Patients with malignancy considered surgically cured are eligible (eg, non- melanoma skin cancer, cancer of the cervix in-situ, ductal carcinoma in situ [Stage 1], Grade 1 endometrial cancer)
* History of unstable or deteriorating cardiac or pulmonary disease within 6 months prior to consent including but not limited to the following:

  * Unstable angina pectoris or myocardial infarction or elective coronary intervention
  * Congestive heart failure requiring hospitalization
  * Uncontrolled clinically significant arrhythmias
  * Symptomatic pulmonary hypertension

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Cohorts A: Proportion of patients with ≥ 20% reduction in red blood cell transfusions over a continuous 12-week treatment period versus baseline red blood cell transfusion history | 12 weeks
  Proportion of patients with ≥ 20% reduction in red blood cell transfusions over a continuous 12-week treatment period versus baseline red blood cell transfusion history
Cohorts B: Proportion of patients with ≥ 20% reduction in red blood cell transfusions over a continuous 12-week treatment period versus baseline red blood cell transfusion history | 12 weeks
  Proportion of patients with ≥ 20% reduction in red blood cell transfusions over a continuous 12-week treatment period versus baseline red blood cell transfusion history
Cohort C: Hemoglobin response rate at Week 12 (increase of ≥ 1.0 g/dL from baseline) | 12 weeks
  Hemoglobin response rate at Week 12 (increase of ≥ 1.0 g/dL from baseline)

SECONDARY OUTCOMES:
Cohort A: Proportion of patients with ≥ 33% reduction in red blood cell transfusion over a continuous 12-week treatment period versus baseline red blood cell transfusion history | 12 weeks
  Proportion of patients with ≥ 33% reduction in red blood cell transfusion over a continuous 12-week treatment period versus baseline red blood cell transfusion history
Cohort B: Proportion of patients with ≥ 33% reduction in red blood cell transfusion over a continuous 12-week treatment period versus baseline red blood cell transfusion history | 12 weeks
  Proportion of patients with ≥ 33% reduction in red blood cell transfusion over a continuous 12-week treatment period versus baseline red blood cell transfusion history
Cohort A: Reduction in red blood cell transfusions over 12 weeks | 12 weeks
  Reduction in red blood cell transfusions over 12 weeks
Cohort A: Reduction in red blood cell transfusions over 24 weeks | 24 weeks
  Reduction in red blood cell transfusions over 24 weeks
Cohort A: Reduction in red blood cell transfusions over 48 weeks | 48 weeks
  Reduction in red blood cell transfusions over 48 weeks
Cohort B: Reduction in red blood cell transfusions over 12 weeks | 12 weeks
  Reduction in red blood cell transfusions over 12 weeks
Cohort B: Reduction in red blood cell transfusions over 24 weeks | 24 weeks
  Reduction in red blood cell transfusions over 24 weeks
Cohort B: Reduction in red blood cell transfusions over 48 weeks | 48 weeks
  Reduction in red blood cell transfusions over 48 weeks
Cohort C: Hemoglobin response rate at Week 24 (increase of ≥ 1.0 g/dL from baseline). | 24 weeks
  Hemoglobin response rate at Week 24 (increase of ≥ 1.0 g/dL from baseline).
Cohort C: Hemoglobin response rate at Week 48 (increase of ≥ 1.0 g/dL from baseline). | 48 weeks
  Hemoglobin response rate at Week 48 (increase of ≥ 1.0 g/dL from baseline).
Change from baseline in hemoglobin over 12 weeks | 12 weeks
  Change from baseline in hemoglobin over 12 weeks
Change from baseline in hemoglobin over 24 weeks | 24 weeks
  Change from baseline in hemoglobin over 24 weeks
Change from baseline in hemoglobin over 48 weeks | 48 weeks
  Change from baseline in hemoglobin over 48 weeks
Changes in serum ferritin levels at 12 weeks versus baseline | 12 weeks
  Changes in serum ferritin levels at 12 weeks versus baseline
Changes in serum ferritin levels at 24 weeks versus baseline | 24 weeks
  Changes in serum ferritin levels at 24 weeks versus baseline
Changes in serum ferritin levels at 48 weeks versus baseline | 48 weeks
  Changes in serum ferritin levels at 48 weeks versus baseline
Changes in liver iron concentration at 48 weeks versus baseline | 48 weeks
  Changes in liver iron concentration at 48 weeks versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (32):
- United States (14):
  - TOI Clinical Research, Cerritos, California
  - [Legal] Children's Hospital Los Angeles, Los Angeles, California
  - University of Californ LA-UCLA, Los Angeles, California
  - UCSF Oakland Benioff ChildHosp, Oakland, California
  - [Legal] Children's Hospital of Orange County on behalf of CHOC Children's Hospital of Orange County, Orange, California
  - UCI Health, Orange, California
  - Children's National Health Hospital, Washington D.C., District of Columbia
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - [Legal] Dr. Vince Clinical Research, LLC and Dr. Vince Clinical Research, P.A., Detroit, Michigan
  - Weill Medical College of Cornell University, New York, New York
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - [Legal] Children's Hospital Medical Center dba Cincinnati Children's, Cincinnati, Ohio
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
- Canada (4):
  - Master Centre for Canada, Mississauga, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - CHU Sainte-Justine Mother and Child University Hospital, Montreal, Quebec
- Egypt (2):
  - Cairo University, Cairo
  - Abu El-Reesh El-Mounira Children University Hospital, Cairo, Egypt
- Italy (4):
  - Galliera Hospital Centro Anemie Congenite, Genova
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - A.O.U. Università Studi della Campania "Luigi Vanvitelli", Naples
  - AORN A. Cardarelli, Napoli
- Lebanon (2):
  - Chronic Care Center, Baabda
  - Hospital Nini, Tripoli
- United Kingdom (6):
  - Sandwell and West Birmingham NHS Trust SCAT/ haematology, Birmingham
  - Barts Health NHS Trust - The Royal London Hospital, London
  - University College Hospital - University College London Hospitals NHS Foundation Trust, London
  - Kings College London, London
  - Hammersmith Hospital - London, London
  - Manchester University NHS Foundation Trust, Manchester